CLINICAL TRIAL: NCT04879550
Title: Prospective Investigation of the Association of Antithrombin III Deficiency With Thrombotic Events in Adult Patients With ECMO
Brief Title: Prospective Investigation of Antithrombin III Deficiency in Adult Patients With ECMO
Status: Completed | Type: Observational
Sponsor: Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Arif Yasin Çakmak, Principal Investigator, Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital
Other Study IDs: HNEAH-KAEK 2019/81-866
Record Dates: First submitted 2021-04-30; First posted 2021-05-10 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Antithrombin III Deficiency; Extracorporeal Membrane Oxygenation Complication
Keywords: Antithrombin III, ECMO
MeSH Terms: conditions — Antithrombin III Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Antithrombin III activity test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- thrombotic event developing / not: Group I: Patients with no bleeding/thrombosis complications Group II: Patients with Thrombotic and/or thromboembolic complications Group III: Patients with bleeding complications
  Interventions: Diagnostic Test: Antithrombin III

INTERVENTIONS:
Diagnostic Test: Antithrombin III — Antithrombin III deficiency causes thrombosis. Is thrombosis in ECMO patients related to Antithrombin III deficiency? Groups with and without thrombosis will be separated and whether it is related to Antithrombin III deficiency will be evaluated.

SUMMARY:
There are publications showing a decrease in Antithrombin III levels of continuous flow and routine heparin therapy in adult patients undergoing Extracorporeal Membrane Oxygenation (ECMO) however, there is not enough data. One of the multifactorial causes affecting bleeding / thrombosis complications and ACT levels may be acquired Antithrombin III deficiency.

The Antithrombin III activity test results from the patients to be included in the study during the study will be recorded immediately after ECMO run, at the 24th hour before the heparin infusion start and at the 48th, 72nd and 96th hours following the follow-up. The results will be analyzed to figure out a relationship between decreasing Antithrombin 3 values and thrombotic events.

DETAILED DESCRIPTION:
ECMO is applied in patients with acute severe heart or lung failure. The treatment protocol of patients undergoing ECMO is carefully arranged against the risk of bleeding / thrombosis.

According to the general protocol, heparin infusion therapy is started at the 24th hour after ECMO application. The risk of bleeding / thrombosis is avoided by adjusting the heparin infusion dose with Activated Clotting Time (ACT) control. However, over time, thrombocytopenia and fluctuations in ACT level are observed in patients. It may be necessary to increase the dose of heparin given during the prolonged period. One of the multifactorial causes affecting bleeding / thrombosis complications and ACT levels may be acquired Antithrombin III deficiency. There are publications reporting a decrease in Antithrombin III levels of continuous flow and routine heparin therapy in adult patients undergoing ECMO; however, there is not enough data.

The Antithrombin III activity test results from the patients to be included in the study during the study will be recorded immediately after ECMO run, at the 24th hour before the heparin infusion start and at the 48th, 72nd and 96th hours following the follow-up. The results will be analyzed to figure out a relationship between decreasing Antithrombin 3 values and thrombotic events.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 18
* Patients with ECMO run for 3 days or more (to be able to determine at least 3 antithrombin 3 levels)

Exclusion Criteria:

* Patients with ECMO run less than 3 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over the age of 18 who underwent ECMO in our hospital are our study population.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Antithrombin 3 activity level | 5 days
  Antithrombin 3 activity test levels will be checked in the first 5 days after ecmo application.

SECONDARY OUTCOMES:
Thrombosis and Bleeding Events | 1 week
  Thrombotic or bleeding complications occurring during ECMO run

CONTACTS AND LOCATIONS:
Overall Officials: Serap AKA, Study Director — Cardiovascular Surgeon
Locations (1):
- Istanbul Dr.Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No